CLINICAL TRIAL: NCT02903836
Title: A Phase II, Randomized, Double-Blind, Multicenter, Comparative Study to Determine the Safety, Tolerability, Pharmacokinetics and Efficacy of Oral Nafithromycin Versus Oral Moxifloxacin in the Treatment of Community-Acquired Bacterial Pneumonia (CABP) in Adults
Brief Title: Phase II Study of Oral Nafithromycin in CABP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: ACM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W-4873-201
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Community-Acquired Bacterial Pneumonia (CABP)
MeSH Terms: interventions — nafithromycin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Nafithromycin 800 mg 3 days (Experimental): PO q24h for 3 days; subjects will receive matching placebo , to maintain the blind
  Interventions: Drug: Nafithromycin 800 mg 3 days
- Nafithromycin 800 mg 5 days (Experimental): PO q24h for 5 days; subjects will receive matching placebo, to maintain the blind
  Interventions: Drug: Nafithromycin 800 mg 5 days
- Moxifloxacin 400 mg (Active Comparator): PO q24h for 7 days;subjects will also receive two nafithromycin placebo tablets PO q24h on Days 1 through Day 7 to maintain the blind
  Interventions: Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: Nafithromycin 800 mg 3 days
  Arms: Nafithromycin 800 mg 3 days
Drug: Nafithromycin 800 mg 5 days
  Arms: Nafithromycin 800 mg 5 days
Drug: Moxifloxacin 400 mg
  Arms: Moxifloxacin 400 mg

SUMMARY:
Study to Determine the Safety, Tolerability, Pharmacokinetics and Efficacy of Oral Nafithromycin Versus Oral Moxifloxacin in the Treatment of Community-Acquired Bacterial Pneumonia (CABP) in Adults

ELIGIBILITY:
Inclusion Criteria:

Meet the clinical criteria for CABP based on following:

1. Clinical symptoms (new or worsening)
2. Vital sign abnormalities
3. Laboratory abnormalities
4. Radiographic evidence of CABP
5. PORT score

Exclusion Criteria:

1. Subjects with any of the following confirmed or suspected types of pneumonia:

   1. Aspiration pneumonia
   2. Hospital-acquired bacterial pneumonia (HABP)
   3. Healthcare-associated bacterial pneumonia (HCAP)
   4. Ventilator-associated bacterial pneumonia (VABP)
   5. Pneumonia that may be caused by pathogen(s) resistant to either study drug
2. Receipt of 1 or more dose(s) of a potentially effective systemic antibacterial treatment for treatment of the current CABP
3. Suspected or confirmed non-infectious causes of pulmonary infiltrates
4. Subjects requiring concomitant adjunctive or additional potentially-effective systemic antibacterial treatment for management of CABP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashima Bhatia, MD PDCR, Study Director — Wockhardt
Locations (6):
- United States (6):
  - A & L Clinical research, Miami, Florida
  - A Plus Research Inc., Miami, Florida
  - RM Medical Research, Inc., Miami, Florida
  - Empire Clinical Research, LLC, Miami Lakes, Florida
  - HCI Metromedic Walkin Medical Center, Bedford, Massachusetts
  - Health Concepts, Bedford, South Dakota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 subjects withdrew consent prior to receiving study drug and 7 subjects whose PK results showed no detectable level of either nafithromycin or moxifloxacin hence 9 subjects excluded from the Safety population.
Groups:
- Nafithromycin 800 mg 3 Days: PO q24h for 3 days; subjects will receive matching placebo , to maintain the blind
  Nafithromycin 800 mg 3 days
- Nafithromycin 800 mg 5 Days: PO q24h for 5 days; subjects will receive matching placebo, to maintain the blind
  Nafithromycin 800 mg 5 days
- Moxifloxacin 400 mg: PO q24h for 7 days;subjects will also receive two nafithromycin placebo tablets PO q24h on Days 1 through Day 7 to maintain the blind
  Moxifloxacin 400 mg
Period: Overall Study
Arm/Group | Nafithromycin 800 mg 3 Days | Nafithromycin 800 mg 5 Days | Moxifloxacin 400 mg
Started | 74 | 73 | 77
Completed | 71 | 69 | 73
Not Completed | 3 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Moxifloxacin 400 mg 7 Days: PO q24h for 7 days;subjects will also receive two nafithromycin placebo tablets PO q24h on Days 1 through Day 7 to maintain the blind
  Moxifloxacin 400 mg 7 days
- Total: Total of all reporting groups
Arm/Group | Nafithromycin 800 mg 3 Days | Nafithromycin 800 mg 5 Days | Moxifloxacin 400 mg 7 Days | Total
Number analyzed (Participants) | 74 | 73 | 77 | 224
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.00 (15.73) | 54.90 (16.90) | 56.10 (15.18) | 56.00 (15.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 35 | 104
  Male | 37 | 41 | 42 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 8 | 13
  Not Hispanic or Latino | 71 | 70 | 68 | 209
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 15 | 18 | 15 | 48
  White | 57 | 52 | 59 | 168
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 8 | 16
  Bulgaria | 14 | 16 | 11 | 41
  Georgia | 8 | 8 | 9 | 25
  Latvia | 4 | 1 | 4 | 9
  Romania | 7 | 4 | 4 | 15
  Serbia | 18 | 19 | 21 | 58
  South Africa | 19 | 21 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response in the ITT Population
Description: The primary efficacy endpoint was clinical response (response, non-response, or indeterminate) at Day 4, tested in the ITT population. Clinical response was determined programmatically using the investigator's assessment of CABP symptoms entered into the eCRF. The severity of the subject CABP symptoms of dyspnea (shortness of breath), cough, production of purulent sputum, and pleuritic chest pain were evaluated on a 4-point scale (absent, mild, moderate, or severe) based upon the CABP Symptom Severity Guidance
Time Frame: Day 4 from start of drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Nafithromycin 800 mg 3 Days | Nafithromycin 800 mg 5 Days | Moxifloxacin 400 mg
Number analyzed (Participants) | 74 | 73 | 77
Participants | 68 | 65 | 67

2. Secondary Outcome: Clinical Response in the Micro-ITT Population
Description: Clinical response (response, non-response, or indeterminate) at Day 4 was also tested in the micro-ITT population as a secondary efficacy endpoint. Clinical response was determined programmatically using the investigator's assessment of CABP symptoms entered into the eCRF. The severity of the subject CABP symptoms of dyspnea (shortness of breath), cough, production of purulent sputum, and pleuritic chest pain were evaluated on a 4-point scale (absent, mild, moderate, or severe) based upon the CABP Symptom Severity Guidance
Time Frame: Day 4 from start of drug administration
Population: The micro-ITT population included all ITT subjects who had at least one baseline Gram-positive or atypical bacterial pathogen known to cause CABP.
Measure: Count of Participants; unit: Participants
Arm/Group | Nafithromycin 800 mg 3 Days | Nafithromycin 800 mg 5 Days | Moxifloxacin 400 mg
Number analyzed (Participants) | 22 | 27 | 20
Participants | 21 | 26 | 18

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent Form to Follow up Visit (Day 31)
Arm/Group | Nafithromycin 800 mg 3 Days | Nafithromycin 800 mg 5 Days | Moxifloxacin 400 mg 7 Days
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/72 | 1/76
Serious Adverse Events (participants affected / at risk) | 1/74 | 1/72 | 2/76
Other Adverse Events (participants affected / at risk) | 11/74 | 9/72 | 6/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nafithromycin 800 mg 3 Days (N=74) | Nafithromycin 800 mg 5 Days (N=72) | Moxifloxacin 400 mg 7 Days (N=76)
Ischemic Stroke (Nervous system disorders) | 0 | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nafithromycin 800 mg 3 Days (N=74) | Nafithromycin 800 mg 5 Days (N=72) | Moxifloxacin 400 mg 7 Days (N=76)
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 3
Hypertension (Vascular disorders) | 3 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT02903836/Prot_SAP_000.pdf